CLINICAL TRIAL: NCT01584505
Title: Randomized, Double-Blind, Active Controlled, 3-Arm Parallel Group, Multi-National, Multi-Centre Study To Evaluate The Cardiac Safety Of Two Doses Of CHF5993 BID Delivered Via HFA PMDI Both Combined With CHF1535 BID Delivered Via HFA PMDI Versus CHF1535 BID Delivered Via HFA PMDI In Patients With Moderate To Severe COPD
Brief Title: Phase II Study to Evaluate the Cardiac Safety of 2 Doses of CHF5993 Both Combined With CHF1535 BID Versus CHF1535 BID in Patients With Moderate to Severe COPD
Acronym: CARSAF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCD-1107-PR-0067; 2011-004759-37 (EudraCT Number)
Record Dates: First submitted 2012-04-23; First posted 2012-04-25 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CHF5993 HFA pMDI dose 1, BID (Experimental): CHF5993 HFA pMDI dose 1, BID
  Interventions: Drug: CHF1535 + CHF5992 dose 1 BID
- CHF5993 HFA pMDI dose 2, BID (Experimental): CHF5993 HFA pMDI dose 2, BID
  Interventions: Drug: CHF1535 + CHF5992 dose2 BID
- CHF1535 HFA pMDI + Placebo (Active Comparator): CHF1535 HFA pMDI BID plus placebo BID
  Interventions: Drug: CHF1535 daily dose

INTERVENTIONS:
Drug: CHF1535 + CHF5992 dose 1 BID — CHF1535 + CHF5992 dose 1 BID for 14 days
  Arms: CHF5993 HFA pMDI dose 1, BID
Drug: CHF1535 + CHF5992 dose2 BID — CHF1535 + CHF5992 dose 2 BID for 14 days
  Arms: CHF5993 HFA pMDI dose 2, BID
Drug: CHF1535 daily dose — CHF1535 daily dose for 14 days
  Arms: CHF1535 HFA pMDI + Placebo

SUMMARY:
Cardiac Safety Study

DETAILED DESCRIPTION:
The purpose of this study is to demonstrate equivalence between CHF1535 plus CHF5992 (two different dosages) over CHF1535 alone in change from baseline in average 24-hour heart rate, as primary end point, and other ECG parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adults ≥ 40years and ≤ 80years old
2. Male subjects: they and/or their partner must be willing to use an approved method of contraception 1) from the time of dose administration and until 30 days after the last dose of study. Subjects must not donate sperm for 30 days after the last dose of study drug
3. Written informed consent obtained by the patient prior to any study related procedures
4. Outpatient with diagnosis of COPD (defined in GOLD guidelines, up to date 2010) at least in the 6 months before the screening visit, including:

   * Smoking history of at least 10 pack years defined as [(number of cigarettes smoked per day) x (number of years of smoking)]/20; both current and ex smokers are eligible. For patients who are in smoking cessation therapy this must be completed at least 1 week before study enrollment
   * Regular use of bronchodilators (e.g. β2-agonist or/and anticholinergics) in the previous 2 months at Visit 0
   * Post-bronchodilator FEV1 ≥ 30% and ≤ 60% of the predicted normal value
   * Post-bronchodilator FEV1/FVC ≤ 0.70

Exclusion Criteria:

1. Pregnant or lactating women or all women physiologically capable of becoming pregnant UNLESS they meet the following definition of postmenopausal: 12 months of natural (spontaneous) amenorrhea or 6 months of spontaneous amenorrhea with already documented serum FSH level > 40mlU/mL or are using one of the following acceptable methods of contraception

   * Surgical sterilization (e.g. bilateral tubal ligation, hysterectomy)
   * Hormonal contraception (implantable, patch, oral)
   * Double-barrier methods (any double combination of: IUD, male or female condom with spermicidal gel, diaphragm, sponge, cervical cap) Reliable contraception should be maintained throughout the study and for 30 days after study drug discontinuation
2. Current diagnosis of asthma or other respiratory disorders (other than COPD) which may interfere with data interpretation according to the investigator's opinion
3. Hospitalization due to COPD exacerbation in the three months prior to screening and during run-in period or COPD exacerbation requiring systemic steroids and or antibiotics in the 6 weeks prior to screening and during run-in period. COPD exacerbation will be defined according to the following criteria: a sustained worsening of the patient condition (dyspnoea, cough and/or sputum production/purulence), from the stable state and beyond normal day-to-day variations, that is acute in onset and necessitates a change in regular medication that includes prescription of oral corticosteroids and/or antibiotics, or need for hospitalization.
4. Patient with COPD who requires regular long term use of oxygen therapy
5. Patient who requires chronic mechanical ventilation for COPD
6. Patient treated regularly with oral or parenteral corticosteroids for their COPD
7. Change of COPD regular medication in the 4 weeks prior to enrollment
8. Unstable CV diseases
9. Known abnormality of any cardiac valve

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2012-04; Primary Completion 2012-09 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in average 24-hour heart rate at Final visit | Day 14 of study treatment
  To assess the effect on change from baseline in average 24h Heart Rate at Day 14 of study treatment

SECONDARY OUTCOMES:
Heart Rate and ECG parameters variation | Day 1 and Day 14 of Study Treatment
  Pre and post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Jörg Kampschulte, MD, Principal Investigator — Arzt für Innere Medizin und Pneumologie, Berlin, Germany
Locations (6):
- Hospital "Lozenets", Sofia, Bulgaria
- Praxis Dr. Kampschulte, Berlin, Germany
- Fővárosi Önkormányzat Szent János Kórháza és Észak-budai Egyesített Kórházai Tüdőgondozó Szakrendelő, Budapest, Hungary
- ISPL Centrum Medyczne Robert M. Mróz, Bialystok, Poland
- State Budgetary Healthcare Institution of Moscow city, Moscow, Russia
- Medicines Evaluation Unit, Langley Building, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Chiesi commits to sharing with qualified scientific and medical Researchers, conducting legitimate research, Patient-level Data, Study-level Data, the Clinical Protocol and the full CSR, providing access to clinical trial information consistently with the principle of safeguarding commercially confidential information and patient privacy. Any shared Patient-level Data is anonymized to protect personally identifiable information.
  Chiesi access criteria and complete process for clinical data sharing is available on the Chiesi Group website.
Access Criteria: Chiesi access criteria and complete process for clinical data sharing is available on the Chiesi Group website.
URL: https://www.chiesi.com/en/chiesi-clinical-trial-data-request-portal/

REFERENCES:
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2011-004759-37
- See also: CSR Synopsis available in the CHIESI Clinical Study Register — https://www.chiesi.com/clinic/CSR_Synopsis_CCD-1107-PR-0067.pdf